CLINICAL TRIAL: NCT02635100
Title: Evaluation of a Multinight (MNT) CPAP Titration Algorithm in Patients With Sleep Apnea.
Brief Title: Multinight CPAP for Sleep Apnea Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI has left the institution
Sponsor: NYU Langone Health (Other)
Collaborators: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-00605
Record Dates: First submitted 2015-12-14; First posted 2015-12-18 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Sleep Apnea; Sleep Disordered Breathing
Keywords: Sleep Disordered Breathing; Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MNT Algorithm (Experimental): All participants will be monitored using an existing (FDA approved) CPAP machine that has been modified to be externally controlled by a computer with the MNT algorithm, for titration.
  Interventions: Other: CPAP machine with MNT algorithm

INTERVENTIONS:
Other: CPAP machine with MNT algorithm — The multinight (MNT) algorithm will be evaluated on patients with Obstructive Sleep Apnea (OSA) over multiple nights while using CPAP in the home for a total of 45 days. In particular the main goal is to assess the behavior of the two main stages of the algorithm:
  1. Fast Track (FT) stage. Assesses if the algorithm reliably and timely reaches approximate therapeutic pressure levels.
  2. Slow Titration (ST) stage.Assesses if data samples are appropriately collected in a pressure range so that the therapeutic pressure can be inferred according to the algorithm proposed.
     1. Five days with standard auto titration.
     2. MNT algorithm : 7 days (maximum) with Fast Track mode, 27 days (maximum) in Slow Titration mode. After PMNT is found, the device remains at PMNT for 5 sessions. Total approximately 45 days.
  Other Names: ICON PLUS

SUMMARY:
Obstructive sleep apnea (OSA) is a prevalent disorders characterized by intermittent obstructions of the upper airway during sleep. Continuous Positive Airway Pressure (CPAP) has been shown to be the most efficacious treatment for OSA. It consists of a small device that provides positive airway pressure delivered by a mask attached to the patients nose/mouth.

DETAILED DESCRIPTION:
The primary purpose of this study is to evaluate the multinight (MNT) algorithm on patients with Obstructive Sleep Apnea (OSA) over 45 nights while using a CPAP machine at home. The researchers are evaluating the performance of the existing algorithm as well as capturing the data to make enhancements.

Two main stages of this algorithm will be assessed:

i. Fast Track (FT) stage. In the FT stage the aim is to assess if the algorithm reliably and timely reaches approximate therapeutic pressure levels.

ii. Slow Titration (ST). In the Slow Titration stage the aim is to assess if data samples have been appropriately collected in a pressure range so that the therapeutic pressure can be inferred according to the algorithm proposed.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* No contradictions to Continuous Positive Airway Pressure (CPAP)
* Able to provide consent

Exclusion Criteria:

° Vulnerable subjects

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Difference in number of residual events between high and low pressure levels | 45 days
  Residual events are represented by a given sleep disordered breathing index SDBIndex
Pressure level obtained during the MNT Fast Track stage | 7 days
Number of days required to reach Fast Track pressure | 7 days
Number of times the algorithm returns to Slow Track from the Fast Track stage | 45 days
Variance in average obstruction of the upper airway during sleep measured by Obstruction Index (OI) | 3 hours
Difference between pressure derived from multinight algorithm (PMNT) and Fast Track pressure | 45 days
Difference between PMNT and sleep lab diagnosed CPAP pressure | 45 days
Number of residual events while using the PMNT function | 45 days

SECONDARY OUTCOMES:
Average comfort rating using CPAP with multinight automated titration | 45 days

CONTACTS AND LOCATIONS:
Overall Officials: David Rapoport, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States